CLINICAL TRIAL: NCT00274365
Title: Consultations in Psychiatry Given to GP's Through Videoconference
Brief Title: Consultations in Psychiatry Through Videoconference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Galil Center for Telemedicine and Medical Informatics (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 4669ctil
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2007-04

CONDITIONS: Remote Consultation [L01.178.847.652.550]
Keywords: general practitioners, psychiatry, videoconference

INTERVENTIONS:
Procedure: videoconference

SUMMARY:
Online consulatations through videoconference in the field of psychiatry given to general practitioners will reduce costs of medical treatment and improve service.

DETAILED DESCRIPTION:
CLINICAL STATE, SATISFACTION AND COST EFFECTIVENESS WILL BE CHECKED DURING 1 YEAR OF ONLINE VIDEO CONFERENCE CONSULTATION TO GENERAL PRACTITIONERS. BPRS, HAMILTON ANXIETY AND DEPRESSION AND CGI SCALES WILL BE COMPLETED.COSTS OF MEDICATIONS, NUMBER OF VISITS, LAB AND OTHER EXAMINATIONS, HOSPITALIZATIONS, MISSING WORKING DAYS WILL BE EVALUATED.

ELIGIBILITY:
Inclusion Criteria:

Referral by general practitioner Age: >18 - Speaking Hebrew or Russion

Exclusion Criteria:

CGI>4 Dementia Drug or alcohol addiction -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Expenditures on medications
No. of visits
Loss of work days
Expenditure on lab tests
Satisfaction
CGI
Hamilton
Somatisation
GHQ11
Q-LES-Q-18
No. of consultations

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Modai, MD, MHA, Study Director — Ruth and Bruce Rappaport Faculty of Medicine, Technion, Haifa, Israel
Locations (1):
- Regional clinic of General Health Services, Hadera, Israel